CLINICAL TRIAL: NCT01296542
Title: A Comparison of Prophylactic Antibacterial Efficacy of Besivance Versus VIGAMOX Administered for Three Days and One Hour Prior to Phacoemulsification
Brief Title: A Comparison of Prophylactic Antibacterial Efficacy of Besivance vs. VIGAMOX Prior to Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bucci Laser Vision Institute (Other)
Responsible Party: Principal Investigator, Frank A. Bucci, Jr., M.D., Principal Investigator, Bucci Laser Vision Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-BV-C
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Results first posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VIGAMOX (Active Comparator): Subjects will self administer drops 4 times daily for 3 days and one drop prior to sample collection
  Interventions: Drug: Moxifloxacin Ophthalmic
- Besivance (Active Comparator): Subjects will self administer drops 4 times daily for 3 days and one drop prior to sample collection
  Interventions: Drug: Besifloxacin Ophthalmic

INTERVENTIONS:
Drug: Moxifloxacin Ophthalmic
  Arms: VIGAMOX
Drug: Besifloxacin Ophthalmic
  Arms: Besivance

SUMMARY:
To compare antibacterial efficacy of Besivance versus VIGAMOX for decreasing bacteria of the conjunctiva and lid margins in cataract patients prior to surgery after both 1 hour and 3 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman 18 years of age or older.
* Physically capable of instilling eye drop or have an appropriate person available to assist in administration of eye drops 4 times a day.
* Scheduled for phacoemulsification with intraocular lens (IOL) implantation for the treatment of cataract.
* Meet the American Society of Anesthesiology (ASA) physical status I, II, or III and be medically cleared for surgery.
* Willing to adhere to the prohibitions and restrictions specified in this protocol.
* Subjects must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* Known allergy or contraindication to the test article(s) or their components.
* Presence of any abnormality or significant illness in the eye that in the investigator's opinion could affect the subject's health or the study parameters.
* Presence of an active ocular infection (bacterial, viral or fungal), or positive history of ocular herpetic infection.
* History of any significant illness that could be expected to interfere with the study parameters. Any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study.
* Use of disallowed therapies (systemic or topical):

  * Fluoroquinolone anti-infective agents (systemic or topical) within 1 week of Visit 1 or anytime after Visit 1 for the duration of the study.
* Use of contact lenses for one week prior to the study and for the duration of the study.
* Received an experimental drug or used an experimental medical device within 21 days before the planned start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank A. Bucci, Jr., MD, Principal Investigator — Bucci Laser Vision Institute
Locations (1):
- Bucci Laser Vision Institute, Wilkes-Barre, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VIGAMOX | Besivance
Started | 30 | 30
Completed | 30 | 28
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VIGAMOX | Besivance | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 7 | 10
  >=65 years | 27 | 23 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Change in Bacterial Colonization of Lid and Conjunctival Cultures After 3 Days
Description: Lid and Conjunctival cultures will be taken to measure bacterial colonization.
Time Frame: Following 3 days of antibiotic drops topically instilled
Measure: Count of Participants; unit: Participants
Arm/Group | VIGAMOX | Besivance
Number analyzed (Participants) | 30 | 28
Participants | 18 | 28

ADVERSE EVENTS:
Arm/Group | VIGAMOX | Besivance
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28
Other Adverse Events (participants affected / at risk) | 0/30 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes